CLINICAL TRIAL: NCT01560689
Title: Open-labeled Trial to Evaluate the Therapeutic Effects of Inhaled BUDESONIDE/FORMOTEROL in Bronchiolitis Obliterans After Allogeneic Stem Cell Transplantation
Brief Title: Inhaled BUDESONIDE/FORMOTEROL in Bronchiolitis Obliterans Following Stem Cell Transplantation
Acronym: alloforb
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Anne Bergeron, MD, PhD, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Bronchiolitis Obliterans; Allogeneic Stem Cell Transplantation
Keywords: bone marrow transplantation; obstructive lung disease; bronchodilators; inhaled steroids; late-onset pulmonary complication
MeSH Terms: conditions — Bronchiolitis Obliterans; Lung Diseases, Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BUDESONIDE/FORMOTEROL (Active Comparator)
  Interventions: Drug: Budesonide/formoterol
- control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide/formoterol — 800 µg/j twice a day, every day
  Other Names: Symbicort
  Arms: BUDESONIDE/FORMOTEROL
Drug: Placebo — Twice a day, every day
  Arms: control

SUMMARY:
The purpose of this study is to determine whether inhaled Budesonide/formoterol is effective in the treatment of bronchiolitis obliterans after allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
Bronchiolitis obliterans (BO) is a life-threatening pulmonary late-onset complication following allogenic stem cell transplantation (SCT), commonly attributed to graft versus host disease (GVHD), and carries a poor prognosis. Although immunosuppressive treatments (IS) represents the main therapeutic approach in this disorder, these medications are rarely efficient and alternative approaches are strongly needed. Because, the combination of inhaled steroids and long-acting bronchodilator are known to decrease respiratory symptoms, prevent exacerbations and improve lung function in chronic obstructive pulmonary diseases with bronchiolar component, they may have beneficial effects in BO. Thus, the investigators conducted a pilot open-labeled trial to evaluate the therapeutic effects of inhaled Budesonide/Formoterol combination (400/12 µg twice a day) without modifying systemic IS received by the patients.

ELIGIBILITY:
Inclusion Criteria:

* adult allogeneic stem cell transplant recipients with clinical respiratory signs assumed to be secondary to BO, without extra-thoracic extensive graft versus host disease

Exclusion Criteria:

* Extensive extra thoracic GVH necessitating increasing immunosuppressive treatments

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
pulmonary function tests | 1 month
Dyspnea based on NYHA classification | 1 month

SECONDARY OUTCOMES:
pulmonary function test | 7 month

CONTACTS AND LOCATIONS:
Overall Officials: bergeron-lafaurie Anne, MD, PhD, Principal Investigator — Pneumology Department, Hopital Saint Louis
Locations (1):
- Hopital Saint Louis APHP, Paris, France